CLINICAL TRIAL: NCT03756012
Title: Multi-Center Evaluation of Clinical Outcomes of Pulse Widths <500 μsec and >1000 μsec During a Temporary Spinal Cord Stimulation Trial
Brief Title: Evaluation of Clinical Outcomes of Pulse Widths in Spinal Cord Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kettering Health Network (Other)
Collaborators: Ohio Pain Clinic (Other)
Responsible Party: Principal Investigator, Amol Soin, Principal Investigator, Kettering Health Network
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Expanded Long Pulse
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Results first posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-02

CONDITIONS: Back Pain; Pain
MeSH Terms: conditions — Back Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Low Pulse Width (<500 μsec) (Active Comparator): Spinal Cord Stimulation System will be programmed to pulse widths <500 μsec.
  Interventions: Device: Algovita Spinal Cord Stimulation System
- High Pulse Width (>1000 μsec) (Active Comparator): Spinal Cord Stimulation System will be programmed to pulse widths >1000 μsec
  Interventions: Device: Algovita Spinal Cord Stimulation System

INTERVENTIONS:
Device: Algovita Spinal Cord Stimulation System — The Algovita™ SCS system is indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with failed back surgery syndrome, intractable low back pain and leg pain.

SUMMARY:
The purpose of this study is to evaluate the effect of pulse widths <500 μsec and >1000 μsec on clinical outcomes during a temporary SCS trial.

DETAILED DESCRIPTION:
The proposed study is a prospective, multi-center, two-arm, randomized, crossover design to be conducted at up to 10 sites. The study will enroll up to 100 subjects in order to include up to 10 subjects in the study per site. Subjects selected to participate in the trial have back and/or leg pain, have been evaluated as a candidate for SCS and have agreed to undergo a temporary SCS trial using the Algovita® system with percutaneous leads. Each subject will be followed during the trial period of approximately 7+/-2 days. The study will end when the last subject has completed the trial period and exited. The expected enrollment period for this study is approximately six months. After exit from the clinical study, subjects will continue to be followed by their physician per usual care. All device and procedure-related AEs will be collected and reported per the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* be eligible for SCS therapy according to the Algovita® SCS system Indications for Use statement
* be undergoing a SCS trial using Algovita® SCS system
* sign a valid, Institutional Review Board (IRB)-approved informed consent form.
* be 18 years of age or older when written informed consent is obtained

Exclusion Criteria:

* be contraindicated for an Algovita® SCS system
* have a cognitive impairment or exhibits any characteristic, that would limit the study candidate's ability to assess pain relief or complete study assessments
* have a life expectancy of less than 2 years
* be participating in another clinical study that would confound data analysis
* have a coexisting pain condition that might confound pain ratings
* have a significant psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio Pain Clinic, Centerville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: patients received both doses
Groups:
- Total Patient Population: This was a case series and all patients received both algorithms; pulse widths <500 µsec and >1000 µsec during a temporary SCS trial with Algovita Trial System. Study ended early and results are only available for total population.
Period: Overall Study
Arm/Group | Total Patient Population
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Patient Population: This was a case series and all patients received both algorithms; pulse widths <500 µsec and >1000 µsec during a temporary SCS trial with Algovita Trial System. Study ended early and results are only available for total population.
  Algovita Spinal Cord Stimulation System: The Algovita™ SCS system is indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with failed back surgery syndrome, intractable low back pain and leg pain.
Arm/Group | Total Patient Population
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 52 [18 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Effect of Pulse Widths on Pain Clinical Outcomes
Description: To evaluate the effect of conventional pulse widths <500 μsec and pulse widths >1000 μsec on clinical outcomes during temporary trial as measured by patient defined pain maps.
Time Frame: For 7 days following intervention
Population: Full statistical analysis did not occur due to premature termination of study. Results were not reported per group, but rather in total since patients received both intervention arms (both pulse widths).
Measure: Count of Participants; unit: Participants
Arm/Group | Total Patient Population
Number analyzed (Participants) | 15
Participants
  Patient subjectively felt coverage was larger with wide pulse width program | 15
  Patient subjectively felt coverage was larger with conventional pulse width program | 0

2. Secondary Outcome: Change in Targeted Pain
Description: To evaluate the effect of conventional pulse widths <500μsecand pulse widths and >1000μsecon clinical outcomes during temporary trial as measured by the number of participants that reported significant change in targeted pain compared to baseline using the NRS at the end of the trial period.
Time Frame: For 7 days following intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Patient Population
Number analyzed (Participants) | 15
Participants
  Patient reported no significant change in pain scores/pain relief | 15
  Patient reported significant change in pain scores/pain relief | 0

3. Secondary Outcome: Distribution of Paesthesia
Description: At end of each arm, subjects will be asked to complete a diagram that shows distribution of paresthesia.
Time Frame: For 7 days following intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Patient Population
Number analyzed (Participants) | 15
Participants
  Larger coverage area with wide pulse width | 15
  Larger coverage area with conventional pulse width | 0

4. Secondary Outcome: Research Participant Program Preference
Description: At the end of the trial period, subjects will be asked to select their favorite program.
Time Frame: For 7 days following intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Patient Population
Number analyzed (Participants) | 15
Participants
  Preferred wide pulse width | 9
  preferred conventional pulse width | 6

5. Secondary Outcome: Quality of Pain Relief
Description: At the end of the trial period, subjects will be asked to rate the quality of the pain relief achieved during the trial (from either arm) using the following ordinal scale; Excellent, Very Good, Good, Fair or Poor
Time Frame: For 7 days following intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Patient Population
Number analyzed (Participants) | 15
Participants
  Excellent | 6
  Very Good | 5
  Good | 4
  Fair | 0
  Poor | 0

6. Secondary Outcome: Research Participant Pain Relief Satisfaction
Description: At the end of the trial period, subjects will be asked to rate their overall satisfaction with the pain relief achieved during the trial (from either arm) using the following ordinal scale; Very Satisfied, Satisfied, Neither Satisfied nor Unsatisfied, Unsatisfied or Very Unsatisfied
Time Frame: For 7 days following intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Patient Population
Number analyzed (Participants) | 15
Participants
  Very Satisfied | 12
  Satisfied | 3
  Neither Satisfied nor Unsatisfied | 0
  Unsatisfied | 0
  Very Unsatisfied | 0

7. Secondary Outcome: ≥ 50% Pain Relief
Description: Number of patients who achieved ≥ 50% pain relief during the trial (from either arm)
Time Frame: For 7 days following intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Patient Population
Number analyzed (Participants) | 15
Participants
  Achieved >/= 50% pain relief during the trial (from either arm) | 15
  Did not achieve >/= 50% pain relief during the trial (from either arm) | 0

8. Secondary Outcome: Rate of AEs
Description: Rate of device-related and/or procedure-related AEs from SCS implant through study completion or study exit.
Time Frame: For 7 days following intervention
Population: was not collected
Arm/Group | Total Patient Population
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 10 days post-implant
Description: Adverse Events were not collected.
Groups:
- Total Patient Population: This was a case series and all patients received both algorithms; pulse widths <500 µsec and >1000 µsec during a temporary SCS trial with Algovita Trial System. Study ended early and results are only available for total population.
  Algovita Spinal Cord Stimulation System: The Algovita™ SCS system is indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with failed back surgery syndrome, intractable low back pain and leg pain.
  Adverse Events were not collected. Study was ended prematurely and results were only provided for total population instead of separate arms since subjects received both interventions.
Arm/Group | Total Patient Population
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT03756012/Prot_SAP_000.pdf